CLINICAL TRIAL: NCT04905173
Title: Comparison of Squat-to-Stand Maneuver With Amyl Nitrite, Valsalva, and Exercise Stress Echocardiography in Inducing Latent Left Ventricular Outflow Obstruction in Hypertrophic Cardiomyopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The decision was made by study team to pursue this as a quality project instead.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey B. Geske, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-003194
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Hypertrophic Cardiomyopathy; Hypertrophic Obstructive Cardiomyopathy; Cardiomyopathy, Hypertrophic
Keywords: squat to stand maneuver; amyl nitrite; echocardiography; valsalva; exercise stress echocardiography; left ventricular outflow tract obstruction; maximal instantaneous gradient; hypertrophic cardiomyopathy; latent obstruction; dynamic obstruction; squat-to-stand
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Ventricular Outflow Obstruction, Left | interventions — Valsalva Maneuver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypertrophic Cardiomyopathy (Experimental): Subjects with a documented diagnosis of hypertrophic cardiomyopathy (HCM) will have an echocardiogram at rest followed by an echocardiogram with Valsalva maneuver as part of regular care. If these tests show no severe obstruction, subjects will continue with both squat-to-stand and amyl nitrite.
  Interventions: Other: Squat-to-stand maneuver; Drug: Amyl nitrite inhalation; Other: Valsalva

INTERVENTIONS:
Other: Squat-to-stand maneuver — Subjects will squat for 5 seconds and then stand. The squat-to-stand exercise will be done up to 10 times, and then immediately undergo echocardiographic imaging.
Drug: Amyl nitrite inhalation — Subjects will inhale amyl nitrite prior to undergoing echocardiographic imaging. This is administered according to current laboratory protocol and is part of standard of care. This is an FDA-regulated drug that will be used as a control and will not be studied experimentally.
Other: Valsalva — Subjects will undergo echocardiographic imaging while performing the Valsalva maneuver. This is according to current laboratory protocol and is part of standard of care.

SUMMARY:
The purpose of this study is to assess the effectiveness of squat-to-stand maneuver in eliciting left ventricular outflow gradients in patients with Hypertrophic Cardiomyopathy (HCM) compared to Valsalva, amyl nitrite inhalation, and exercise stress echocardiogram (ESE).

DETAILED DESCRIPTION:
Left ventricular hypertrophy and abnormal ventricular configuration result in dynamic left ventricular outflow obstruction in ~75% of HCM patients, which is associated with increased cardiac morbidity and mortality. However, the dynamic nature of the gradient can make obstruction difficult to identify. Provocative maneuvers such as Valsalva maneuver, administration of amyl nitrite, and ESE are currently used to assess for obstruction.

A shortage of amyl nitrite beginning in December 2018 spurred a search for alternative provocative maneuvers. Beginning in February 2019, the Mayo Clinic echocardiography laboratory began utilizing a squat-to-stand maneuver as an alternative to amyl nitrite inhalation. Anecdotally, the squat-to-stand maneuver, which decreases both preload and afterload, has been successful in provoking latent left ventricular outflow obstruction. A retrospective study (Peng et al, in progress) studying 119 patients who performed the squat-to-stand maneuver between February and September 2019 demonstrated squat-to-stand to be a more robust provocative maneuver than the Valsalva maneuver for identifying severe dynamic left ventricular obstruction with Doppler echocardiography. Squat-to-stand elicited latent obstruction in a greater proportion of the study participants and higher average gradients. It also demonstrated the potential to alter clinical management - six patients had severe obstruction only with squat-to-stand (otherwise would not have been diagnosed) and subsequently underwent septal reduction surgery.

The recent return of amyl nitrite to the echocardiography laboratory creates an opportunity for direct comparison with squat-to-stand, particularly regarding cost savings and diagnostic performance. The primary purpose of this study is to evaluate the efficacy and degree of provocation of left ventricular outflow gradients by the squat-to-stand maneuver compared to amyl nitrite inhalation in patients with HCM undergoing echocardiography. Squat-to-stand will also be compared with other provocation methods, including Valsalva maneuver, which should be performed on every patient going on to squat-to-stand, and ESE when available. Validating this novel provocative maneuver can broaden the toolbox of techniques used to elicit left ventricular outflow gradients and improve clinical evaluation and management of symptomatic HCM patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 y/o referred for an outpatient echocardiogram.
* Clinical diagnosis of Hypertrophic Cardiomyopathy (HCM).
* Both amyl nitrite inhalation and squat-to-stand maneuver performed during echocardiogram.

Exclusion Criteria:

* Patients < 18 at the time of echocardiogram.
* Studies without documented provocative maneuvers.
* Patients with resting obstruction (MIG > 50 mmHg).
* Patients unable to undergo the squat-to-stand as protocolled based because of physical limitations.
* Patient with contraindications to amyl nitrite administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Severe provokable obstruction | Baseline
  Percentage of patients with provokable obstruction (rest gradient < 30 mmHg AND gradient w/ maneuver ≥ 30 mmHg) by provocation technique

SECONDARY OUTCOMES:
Maximal instantaneous gradient | Baseline
  Maximal instantaneous gradient (MIG) by provocation technique measured in mm Hg
Completion of squat-to-stand maneuver | Baseline
  Percentage of patients unable to complete a squat-to-stand maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Geske, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials